CLINICAL TRIAL: NCT06929247
Title: Clinical and Radiographic Evaluation of Pulpotomy Using Neoputty MTA Versus Pulpectomy Using Metapex in Vital Primary Molars Diagnosed With Symptomatic Irreversible Pulpitis in Children Aged 4 to 9 Years: A Randomized Controlled Trial
Brief Title: Clinical and Radiographic Evaluation of Pulpotomy Using Neoputty MTA Versus Pulpectomy Using Metapex in Vital Primary Molars Diagnosed With Symptomatic Irreversible Pulpitis in Children Aged 4 to 9 Years.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Nashaat Mohamed (Other)
Responsible Party: Sponsor-Investigator, Mohamed Nashaat Mohamed, assistant lecture, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230730
Record Dates: First submitted 2025-04-04; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pulpitis - Irreversible
MeSH Terms: interventions — Pemetrexed; Calcium Hydroxide; iodoform

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of trial participants or clinical investigators will not be possible due to evident differences between the two trial interventions. However, postoperative clinical outcomes will be assessed by an experienced pediatric dentist who is blinded to the treatment allocation, while the radiographic outcomes will be independently assessed by two different pediatric dentists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulpotomy (Experimental): Pulpotomy using Neoputty Mineral Trioxide Aggregate
  Interventions: Procedure: Pulpotomy using Neoputty Mineral Trioxide Aggregate
- pulpectomy (Active Comparator): Single-visit pulpectomy using Metapex
  Interventions: Procedure: single visit pulpectomy using metapex

INTERVENTIONS:
Procedure: Pulpotomy using Neoputty Mineral Trioxide Aggregate — Pulpotomy (Test Group): Removal of coronal pulp followed by Neoputty MTA placement and restoration.
  Other Names: MTA
  Arms: Pulpotomy
Procedure: single visit pulpectomy using metapex — pulpectomy: removal of radicular pulp followed by metapex placement and final restoration
  Other Names: calcium hydroxide with iodoform
  Arms: pulpectomy

SUMMARY:
itle: Evaluation of Pulpotomy using Neoputty MTA vs. Pulpectomy using Metapex in Children (4-9 years).

Objective: Compare clinical and radiographic success of pulpotomy vs. pulpectomy for vital primary molars with irreversible pulpitis.

Design: Randomized controlled trial with 2-arm parallel groups.

Participants: Healthy children aged 4-9 with specific inclusion/exclusion criteria.

Outcomes: Primary (pain relief, absence of complications) and secondary (radiographic success).

DETAILED DESCRIPTION:
Background and Rationale Treating irreversible pulpitis in primary molars is challenging due to complex root canal anatomy and rapid progression of pulp inflammation. Pulpectomy is the standard approach, but its technical difficulty often necessitates referral to specialists. New bioactive materials like Neoputty MTA and improved understanding of pulp biology justify reevaluation of less invasive treatments like pulpotomy. This study addresses the lack of clinical trials comparing pulpotomy with pulpectomy in cases of irreversible pulpitis in primary molars. Aim To compare the clinical and radiographic success of pulpotomy using Neoputty MTA vs. pulpectomy using Metapex in vital primary molars with symptomatic irreversible pulpitis in children aged 49 years. Hypothesis Null Hypothesis: No significant difference in treatment outcome between pulpotomy and pulpectomy.

Methodology Participants

* Setting: Pediatric Dentistry Department, Faculty of Dentistry, Cairo University
* Eligibility: Healthy (ASA I/II), cooperative children aged 49 with vital primary molars exhibiting signs of irreversible pulpitis.
* Exclusion: Necrotic pulp, periapical pathology, pathological mobility, poor restorability, or refusal of crown placement. Sample Size 40 teeth per group (total 80), accounting for 15% dropout. Based on expected 20% difference in outcomes and 80% power. Interventions Pulpotomy (Test Group): Removal of coronal pulp followed by Neoputty MTA placement and restoration. Pulpectomy (Control Group): Complete root canal debridement and obturation with Metapex. Same restoration and crown protocol. Outcomes Primary: Post-operative pain (VAS), clinical and radiographic success over 12 months.

Secondary: Pain assessment at 24 hours and 7 days post-treatment using VAS. Follow-up Timeline Evaluations at baseline, 24h, 1w, 3m, 6m, 9m, and 12m post-intervention. Randomization and Blinding Randomization via opaque sealed envelopes. Outcome assessors blinded.

ELIGIBILITY:
Inclusion Criteria:

* 1. Symptoms typical of irreversible pulpitis, such as spontaneous, unprovoked pain lasting from a few seconds to several hours prior to the dental visit, or pain exacerbated by hot and/or cold stimuli that lingers even after the stimuli are removed.

  2. Confirmation of tooth vitality post-deroofing the pulp chamber, indicated by the presence of uniformly reddish-pink vascular tissue (healthy pulp) upon visual inspection of pulpal hemorrhage.

  3. Confirmation of radicular pulp health post-coronal pulp amputation, demonstrated by achieving radicular pulp hemostasis within 8 minutes using a 5% sodium hypochlorite (NaOCl)-dampened cotton pellet.

  4. The primary molar must be restorable with a stainless-steel crown. 5. Any physiological root resorption present must be less than one-third of the normal root length.

Exclusion Criteria:

* 1. Clinical signs of pulpal infection, such as pathologic tooth mobility, parulis/fistula, or soft tissue swelling.

  2. Pre-operative periapical radiographs indicating furcal radiolucency extending more than half the distance from the furcation to the periapical area.

  3. Pre-operative periapical radiographs showing periapical radiolucency. 4. Pre-operative periapical radiographs indicating pathological root resorption.

  5. Signs of necrosis in pulp tissue post-deroofing, such as avascular or minimally bleeding pulp, or yellowish necrotic areas/purulent exudate.

  6. Evidence of extensive radicular pulp inflammation post-coronal pulp amputation, indicated by bleeding that continues after 8 minutes of compression with a NaOCl-soaked cotton pellet.

  7. Parents unwilling to place full coverage crowns post-treatment. 8. If both primary molars in the quadrant are painful and the clinical diagnosis of irreversible pulpitis between the teeth is not sharply defined.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | after 24h , 1week, 3 months, 6 months ,9 months and 12 months
  by Visual analog scale from zero to ten. which zero is better outcome and ten is worse outcome

SECONDARY OUTCOMES:
Pain on percussion | after 24h , 1week, 3 months, 6 months ,9 months and 12 months
  Tapping the tooth with the blunt end of the mirror
Number of tooth with Swelling or fistula | after 24h , 1week, 3 months, 6 months ,9 months and 12 months
  Clinical examination
Mobility | after 24h , 1week, 3 months, 6 months ,9 months and 12 months
  Clinical examination
Radiolucency at the furcation or periapical area | after 24h , 1week, 3 months, 6 months ,9 months and 12 months
  Digital periapical intraoral radiograph
Internal or external root resorption | after 24h , 1week, 3 months, 6 months ,9 months and 12 months
  Digital periapical intraoral radiograph